CLINICAL TRIAL: NCT01814995
Title: Combining Motivational Support, Meal Preparation Training, and a Tapering Course of Meal Replacements To Achieve Vascular Risk Reduction in Women With a Gestational Diabetes History (MoMM)
Brief Title: Motivational Support and Meal Preparation Training to Reduce Vascular Risk After Gestational Diabetes
Acronym: MoMM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Kaberi Dasgupta, MD, MSc, FRCP (C), Associate Professor, McGill University, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CIHR-CAI117789
Record Dates: First submitted 2013-03-18; First posted 2013-03-20 (Estimated); Last update posted 2014-09-11 (Estimated); Status verified 2014-09

CONDITIONS: Gestational Diabetes Mellitus With Baby Delivered
Keywords: behavioural; diabetes prevention; overweight; physical activity; gestational diabetes
MeSH Terms: conditions — Overweight; Motor Activity; Diabetes, Gestational | interventions — Nutritional Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nutrition/Physical Activity Intervention (Experimental): There will be four in-person group sessions (1/month), two including the participants' partners, and all with on-site child care. Sessions will include preparation of a healthy meal (hands-on) and discussions of mindful eating, balanced meals, portion sizes, and preparing food at home, under a dietitian's supervision. Sessions will also include a one-hour physical activity information/practice session with a kinesiologist. Participants will track daily step counts with a pedometer and aim to eventually reach more than 10,000 steps/day. They will also receive instruction and demonstration from a kinesiologist of some simple resistance exercises they may perform at home. Between sessions, participants will receive advice and support through a study-specific website and telephone calls.
  Interventions: Behavioral: Nutrition/Physical Activity Intervention

INTERVENTIONS:
Behavioral: Nutrition/Physical Activity Intervention — Please see Arm description.
  Other Names: Lifestyle Intervention; Diabetes Prevention Intervention

SUMMARY:
Women with a history of 'diabetes in pregnancy' or Gestational Diabetes (GDM) have a high risk for type 2 diabetes later in life. This can often be prevented, however, with improvements in eating habits and higher physical activity levels. However, many women find it difficult to alter their lifestyle habits, especially if they have young children. In adults with type 2 diabetes, the investigators have been studying the effects of combining nutrition education with meal preparation training and pedometer-based self-monitoring to improve eating habits and increase activity levels. The investigators have shown that such a strategy can reduce hemoglobin A1C by 0.3% and correlates with small reductions in weight (Dasgupta et al, International Journal of Behavioural Nutrition and Physical Activity, 2012). In developing the present interventional study, we presented this strategy to women with a GDM history and asked them how they would modify it to suit their needs. They expressed strong interest in such an approach but emphasized a need to involve their spouses and provide childcare support. They did not express interest in use of meal replacements. Therefore, in MoMM-intervention phase, the investigators will examine the effects of a once per month (4 session) program combined with Internet/telephone-based support. The four sessions with include meal preparation training, strategies to limit mindless eating and improve meal content and portion control. All sessions will offer child care. Two sessions will involve spouses. The investigators will assess effects on weight, BMI, DXA measures of fat, and measures of insulin resistance and blood pressure. This single-arm intervention study may lead ultimately to a randomized controlled trial.

DETAILED DESCRIPTION:
The investigators have adopted a single-arm intervention pilot study to assess the potential effects of a nutrition/physical activity behavioural intervention in women with a history of GDM within the past 5 years. The investigators have designed the intervention to include in-person sessions- but at a feasible frequency for busy mothers- as well as telephone calls and an on-line discussion forum, to provide an ongoing source of support, information, and accountability. Further, participants' partners will be invited to some of the in-person sessions and childcare will be provided on-site. Importantly, there are no meal replacements included, despite the study title, because focus group discussions indicated that this was not of interest to the target population.

The investigators will hold in-person sessions at a frequency of once per month over a 4-month period. In addition to the in-person, on-site sessions, we will arrange for participants to have in a grocery store 'tour' led by a student from the McGill School of Dietetics and Human Nutrition BSc program. This will allow a review of label reading and interpretation as well as tips on produce selection. Details of the intervention are provided under the trial arm section below.

ELIGIBILITY:
Inclusion Criteria:

1. Prior history of GDM
2. Body mass index (BMI) ≥ 24 kg/m2
3. Ability to speak and read English or French

Exclusion Criteria:

1. Type 1 diabetes
2. Type 2 diabetes
3. Use of antihyperglycemic medication
4. Pregnant or planning to become pregnant again in the next year
5. Food allergies
6. Chronic condition/ medications that could impact weight (e.g. malignancy, weight loss medications, anti-depressants)
7. Current smoker

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2012-01; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
percentage change in weight in participant | 16 to 20 weeks
  Women with a GDM history within the past 5 years are enrolled with a BMI at or above 24 kg/m2. Weight will be measured to the nearest 0.1 kilogram with an automated scale. We will subtract the post intervention weight from the baseline weight to compute the change in weight. We will divide this value by the baseline weight to compute the percentage change in weight from baseline.

SECONDARY OUTCOMES:
change in BMI | 16 to 20 weeks
  We will subtract the baseline BMI from the post intervention BMI of the participant. For computation of the BMI values, weight is divided by the square of the height. The latter is assessed with the aid of a stadiometer.
change in waist circumference | 16 to 20 weeks
  Waist circumference will be measured midway between the iliac crest and the lower rib margin. We will subtract the baseline value from the post intervention value to compute the change in waist circumference.
change in waist to hip ratio | 16 to 20 weeks
  Hip circumference will be measured at the point of greatest posterior extension of the buttocks. Waist to hip ratio will be computed (waist in cm divided by height in cm). The baseline waist to hip ratio will be subtracted from the post intervention waist to hip ratio for computation of the change in waist to hip ratio.
change in total body fat | 16 to 20 weeks
  We will perform Dual-Energy X-ray absorptiometry measurements of total body composition (soft lean tissue, bone mineral and fat mass)to estimate the percentage of total body fat content of subjects. We will subtract baseline total body fat from post intervention total body fat to compute change in total body fat.
adbominal adiposity | 16 to 20 weeks
  Using DXA measures, we will estimate abdominal adiposity and subtract baseline from post intervention values.
change in fasting glucose levels | 16 to 20 weeks
  Following an overnight fast, venous blood will be sampled for assessment of fasting glucose. Baseline values will be subtracted from final values for computation of change in fasting glucose levels.
change in 1-hour glucose level following 75-gram glucose load | 16 to 20 weeks
  Following acquistion of fasting venous blood samples, participants will ingest a 75 gram glucose solution. Venous blood will again be sampled for glucose level measurement. We will subtract the baseline 1-hour glucose value from the post intervention 1-hour glucose value to compute change in 1-hour glucose level following 75- gram glucose load. The 60-minute glucose value following the 75-gram glucose load has been demonstrated to be a good predictor of future development of diabetes among those with a normal fasting glucose level.
Proportion with elevated 1-hour glucose level following 75-gram glucose load | 16 to 20 weeks
  Following acquistion of fasting venous blood samples, participants will ingest a 75 gram glucose solution. Venous blood will again be sampled for glucose level measurement. The 60-minute glucose value following the 75-gram glucose load has been demonstrated to be a good predictor of future development of diabetes among those with a normal fasting glucose level (i.e., higher risk with glucose values above 8.6 mmol/L). We will calculate the proportion of participants will a 1- hour glucose level above 8.6 mmol/L at baseline and post intervention and will compare these proportions.
change in 2-hour glucose level following 75-gram glucose load | 16 to 20 weeks
  Following acquistion of fasting venous blood samples, participants will ingest a 75 gram glucose solution. Venous blood will again be sampled for glucose level measurement at 1 hour and at 2 hours after ingestion. We will subtract the baseline 2-hour glucose value from the post intervention 2-hour glucose value to compute change in 2-hour glucose level following 75- gram glucose load.
change in fasting insulin levels | 16 to 20 weeks
  Following an overnight fast, venous blood will be sampled for assessment of fasting insulin. Baseline values will be subtracted from final values for computation of change in fasting insulin levels.
change in 1-hour insulin level following 75-gram glucose load | 16 to 20 weeks
  Following acquistion of fasting venous blood samples, participants will ingest a 75 gram glucose solution. Venous blood will again be sampled for insulin level measurement. We will subtract the baseline 1-hour insulin value from the post intervention 1-hour insulin value to compute change in 1-hour insulin level following 75- gram glucose load.
change in 2-hour insulin level following 75-gram glucose load | 16 to 20 weeks
  Following acquistion of fasting venous blood samples, participants will ingest a 75 gram glucose solution. Venous blood will again be sampled for insulin level measurement at 1 hour and at 2 hours after ingestion. We will subtract the baseline 2-hour insulin value from the post intervention 2-hour insulin value to compute change in 2-hour insulin level following 75- gram glucose load.
change in Homeostatic Model Assessment of insulin resistance (HOMA-IR) | 16 to 20 weeks
  We will use fasting glucose and insulin values to compute a measure of insulin resistance, the Homeostatic Model Assessment (HOMA) [Fasting insulin (microunits/mL) X fasting glucose (mmol/L) divided by 22.5]. We will subtract the baseline value from the post intervention value to compute the change in HOMA-IR.
change in insulin sensitivity index 0, 120 (ISI) | 16 to 20 weeks
  Using the ratio of the serum insulin levels at the 0 minute and 120-minute time points, the insulin sensitivity index (ISI 0, 120), another marker of insulin resistance, will be calculated as proposed in Gutt M, Davis CL, Spitzer SB, Llabre MM, Kumar M, Czarnecki EM et al. Validation of the insulin sensitivity index (ISI(0,120)): comparison with other measures. Diabetes Res Clin Pract 2000; 47(3):177-184. We will subtract the ISI 0,120 value at baseline from the post intervention value to compute the change in ISI 0,120.
change in systolic blood pressure | 16 to 20 weeks
  Systolic blood pressure will assessed with the participant seated in a quiet room with the arm supported. Measurements will be taken with an automated device at 1-minute intervals for 6 sequential measurements. The latter 5 measurements will be averaged. The baseline (average) systolic blood pressure will be subtracted from the post intervention (average) systolic blood pressure for computation of the change in systolic blood pressure.
change in diastolic blood pressure | 16 to 20 weeks
  Diastolic blood pressure will assessed with the participant seated in a quiet room with the arm supported. Measurements will be taken with an automated device at 1-minute intervals for 6 sequential measurements. The latter 5 measurements will be averaged. The baseline (average) diastolic blood pressure will be subtracted from the post intervention (average) diastolic blood pressure for computation of the change in systolic blood pressure.
change in daily step count | 16 to 20 weeks
  Step counts will be computed at baseline and post intervention assessments using a Yamax SW-200 pedometer, based on one week of recording. The mean daily step count will be computed. The change in average daily step count will be calculated by subtracting the baseline value from the final value.
change in physical activity level | 16 to 20 weeks
  Participants will wear an accelerometer (AGGT3X-Plus 512MB GT3X-Plus Triaxial Activity Monitor) at the hip (elastic belt provided) for a 7-day period at baseline and post intervention. From accelerometry data, we will calculate mean sedentary time per day as well as time at light, moderate, and vigorous activity levels. We will compute changes in mean daily time at various activity levels by subtracting baseline from post intervention values.
change in total cholesterol | 16 to 20 weeks
  Total cholesterol will be measured using spectrophotometer at baseline and post intervention. The baseline value will be subtract from the post intervention value.
change in high density lipoprotein cholesterol | 16 to 20 weeks
  High density lipoprotein cholesterol will be measured using spectrophotometer at baseline and post intervention. The baseline value will be subtract from the post intervention value.
Change in triglyceride levels | 16 to 20 weeks
  Triglyceride levels will be measured using spectrophotometer at baseline and post intervention. The baseline value will be subtract from the post intervention value.
change in low density lipoprotein cholesterol | 16 to 20 weeks
  The low density lipoprotein cholesterol will be calculated using the Friedewald equation at baseline and post intervention, based on total cholesterol and high density lipoprotein cholesterol values measured using spectrophotometer. The baseline values will be subtracted from post intervention values.
change in total cholesterol to high density lipoprotein cholesterol ratio | 16 to 20 weeks
  Total cholesterol and high density lipoprotein cholesterol will be measured using spectrophotometer at baseline and post intervetion; the total cholesterol to high density lipoprotein cholesterol ratio will be computed at both of these time points. The change in this ratio will be computed by subtracting the baseline ratio from the post intervention ratio.
change in weight of participant's spouse | 16 to 20 weeks
  We will subtract the post intervention weight from the baseline weight to compute the change in weight (participant report). We will divide this value by the baseline weight to compute the percentage change in weight from baseline.
Change in eating habits | 16 to 20 weeks
  We will use the nutritional measures interview from the baseline and post-intervention assessments; we will use the food groups estimation (for both fruits and vegetables separately and combined, as well as Meat and Alternatives, Milk and Alternatives, Grains products) by portions, the water intake estimation in mL, the energy in kcal in the 24 hour recall at both of these time points and subtract the baseline values from the post intervention values.
Change in eating outside of the home | 16 to 20 weeks
  During the baseline and the post-intervention interviews, we will be asking the participants how many times, on average, they eat outside of the home per month. We will subtract the post-intervention value from the baseline value to see the change in eating out.
Change in cooking ability | 16 to 20 weeks
  During the baseline and post-intervention assessments, we ask them about their ability to cook from basic ingredients. We have given a value from 1-7 for the responses to this question, and will calculate the change in this value by subtracting the post-intervention response from the baseline response.
Change in fiber intake | 16 to 20 weeks
  Using the eaTRACKER.ca website to track participant food intake, we will take the average of the first month's fiber intake to the last month's fiber intake and subtract the first month average to the last month average to determine the change.
Change in anxiety and depression | 16-20 weeks
  Using the "Hospital Anxiety and Depression scale" (HADS), Zigmond & Snaith, 1983, we will score the participant responses (a total of 21 for anxiety and a total of 21 for depression), during both the baseline and the post-intervention assessments. We will then subtract the baseline values from the post-intervention values to calculate the change in anxiety and depression.
Change in measure of self-efficacy for eating control | 16-20 weeks
  The Weight Efficacy Life-Style Questionnaire (WEL) will be used during baseline and the post-intervention assessments. We will then use the methods outlined (Clark et al., 1991) to yield 5 sub-scale scores that measure "negative emotions (e.g., eating when sad or anxious), availability (e.g., eating when food is readily available, such as at a party), social pressure (e.g., declining food when others are encouraging eating), physical discomfort (e.g., eating when fatigued or in pain), and positive activities (e.g., eating when watching TV or reading)" (Dutton, GR, et al. 2004). The baseline values will be subtracted from the post-intervention values to yield the change.
Change in perceived stress | 16 to 20 weeks
  Using the perceived stress scale questionnaire (Cohen, S. and Williamson, G. Perceived Stress in a Probability Sample of the United States, 1988.), we will score the responses from the participants at the baseline and post-intervention assessments and calculate the change by subtracting the score of the baseline assessment from the post-intervention assessment.
Change in reported physical activity | 16 to 20 weeks
  Using the "International Physical Activity Questionnaire", we will assess the change from the baseline and post-intervention reported physical activity. We will score the responses using the methods outlined for this questionnaire (http://www.ipaq.ki.se/scoring.htm) and subtract the baseline score from the post-intervention score to report the change.
Change in mindful eating | 16 to 20 weeks
  During the baseline and the post-intervention assessments, we will be using the "mindful eating questionnaire (MEQ)" (Framson, C., et al , 2009), to measure mindful eating. The change will be calculated by subtracting the baseline scores from the post-intervention scores.

CONTACTS AND LOCATIONS:
Overall Officials: Kaberi Dasgupta, MD, MSc, Principal Investigator — McGill University and McGill University Health Centre
Locations (2):
- Canada (2):
  - McGill University Health Centre, Montreal, Quebec
  - Sir Mortimer Davis Jewish General Hospital, Montreal, Quebec

REFERENCES:
- [Background] Dasgupta K, Da Costa D, Pillay S, De Civita M, Gougeon R, Leong A, Bacon S, Stotland S, Chetty VT, Garfield N, Majdan A, Meltzer S. Strategies to optimize participation in diabetes prevention programs following gestational diabetes: a focus group study. PLoS One. 2013 Jul 4;8(7):e67878. doi: 10.1371/journal.pone.0067878. Print 2013. PMID 23861824
- [Background] Leong A, Rahme E, Dasgupta K. Spousal diabetes as a diabetes risk factor: a systematic review and meta-analysis. BMC Med. 2014 Jan 24;12:12. doi: 10.1186/1741-7015-12-12. PMID 24460622
- [Result] Brazeau AS, Leong A, Meltzer SJ, Cruz R, DaCosta D, Hendrickson-Nelson M, Joseph L, Dasgupta K; MoMM study group. Group-based activities with on-site childcare and online support improve glucose tolerance in women within 5 years of gestational diabetes pregnancy. Cardiovasc Diabetol. 2014 Jun 30;13:104. doi: 10.1186/1475-2840-13-104. PMID 24981579
- See also: Main results — http://www.cardiab.com/content/13/1/104
- See also: related systematic review (spousal diabetes concordance) — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC3900990/
- See also: Focus group study that informed intervention design — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC3701629/